CLINICAL TRIAL: NCT01237496
Title: Longitudinal Analysis of HBV-specific T Cell Responses in Patients With HBeAg-negative Chronic Hepatitis B (CHB) Treated With Pegylated Interferon Alfa-2a (40 KD) (Pegasys - RO258310). Immunology Sub-study of ML18253
Brief Title: Analysis of HBV-Specific Immune Response in Patients With HBeAg Negative Chronic Hepatitis B Treated With Pegasys (Peginterferon Alfa-2a (40KD)) - Immunology Sub-Study of ML18253
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18675
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly

SUMMARY:
This study will evaluate immune responses in patients with HBeAg-negative chronic Hepatitis B treated with Pegasys (peginterferon alfa-2a). Eligible patients will have been randomized in study ML18253 to receive Pegasys 180 mcg subcutaneously for 48 or 96 weeks. Sample collection period for each patients will occur in the first 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-55 years of age
* Chronic HBeAg negative hepatitis B
* Liver disease consistent with chronic hepatitis documented by liver biopsy within 18 months prior to enrollment
* Participation in study ML18253.

Exclusion Criteria:

* Interferon-based or any systemic anti-HBV therapy </= 12 months prior to first dose of study drug
* Antiviral, anti-neoplastic, or immunomodulatory treatment </= 12 months prior to first dose of study drug
* Nonresponders to previous interferon therapy and resistant to lamivudine
* Co-infection with hepatitis A, C or D, or with human immunodeficiency virus (HIV)
* Hepatocellular cancer
* Compensated (Child A, score 6) or decompensated liver disease (Child B or C)
* History or evidence of medical condition associated with chronic liver disease other than HBV

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
CD4 and CD8 mediated immune response: Interferon-y (ELISPOT analysis, flow cytometry) | 24 weeks
CD4 and CD8 mediated immune response: Interleukin-2 production (Flow cytometry) | 24 weeks
CD4 and CD8 mediated immune response: Cytokine profile analysis by supernatant culture | 24 weeks
CD4 and CD8 mediated immune response: Proliferative response upon T-cell stimulation | 24 weeks
CD8 response in HLA-A2 positive patients | 24 weeks

SECONDARY OUTCOMES:
Profile of proinflammatory cytokines: analysis of cytokines in serum | 24 weeks
HBV viremia (HBV RNA assessed by COBAS PaqMan HCV test) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (5):
- Italy (5):
  - Bologna
  - Brescia
  - Milan
  - Parma
  - Reggio Emilia